CLINICAL TRIAL: NCT00367016
Title: Immunologic Basis of Anti-IgE Therapy (Study II: On Patients With Asthma)
Acronym: Xolair
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 200312064
Record Dates: First submitted 2006-08-19; First posted 2006-08-22 (Estimated); Results first posted 2021-07-13 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-06

CONDITIONS: Asthma; Allergic Rhinitis; Atopic Dermatitis
MeSH Terms: conditions — Asthma; Rhinitis, Allergic; Dermatitis, Atopic | interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omalizumab (Experimental): Subjects will receive subcutaneous Omalizumab for 6 months. Prior to Omalizumab administration, all subjects will undergo screening studies, including spirometry, blood test and skin test. Blood test includes comprehensive metabolic panel, CBC, and total and free IgE levels. Skin test will be done with a panel of 7 common allergens
  Interventions: Drug: Omalizumab
- Placebo (Experimental): Subjects will receive subcutaneous placebo for 6 months. Prior to placebo administration, all subjects will undergo screening studies, including spirometry, blood test and skin test. Blood test includes comprehensive metabolic panel, CBC, and total and free IgE levels. Skin test will be done with a panel of 7 common allergens
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Omalizumab — Xolair (Omalizumab) will be given by subcutaneous injection according to Ige level and weight calculation.
  Other Names: Xolair
  Arms: Omalizumab
Drug: Placebo — Placebo, given by subcutaneous injection.
  Arms: Placebo

SUMMARY:
The purpose of this study is to look at measures that will help scientists understand the way Omalizumab, an FDA-approved anti-allergy medication, works.

DETAILED DESCRIPTION:
IgE is a key molecule involved in immediate hypersensitivity and plays a major role in the pathogenesis of allergic diseases. Recently, a therapy based on the use of anti-IgE antibody has been developed by a pharmaceutical company, Genentech. A number of clinical trials have demonstrated that these antibodies are efficacious in treatment of allergies, including allergic rhinitis and asthma. The medication Omalizumab (Xolair) has recently been approved by the FDA for treatment of asthma.

The mechanism underlying the beneficial effect of this therapy is not completely understood, but is likely to be related to the marked reduction in the IgE level. Of note is the concomitant accumulation of IgE-anti-IgE complexes in the sera. Another remarkable effect of the treatment is the substantial reduction in the FcεRI level on basophils, which is likely a key factor contributing to the therapeutic benefit of the drug. The existing literature suggests that the reduction in the IgE level is likely to result in a down-regulation of another IgE receptor, FcεRII/CD23. Because of the known immunomodulatory function of FcεRII, anti-IgE therapy may result in alterations of the immune system, in addition to simple absorption of IgE.

We propose to conduct mechanistic studies of anti-IgE therapy. The objectives are to address how anti-IgE therapy works and how it might affect the immune system in general. The proposed studies also take advantage of this well-defined therapy to address some basic questions regarding the immune system. Our hypothesis is that anti-IgE therapy may have general effects on the immune system, such as reduced IgE-mediated antigen presentation by antigen-presenting cells and suppressed allergen-specific IgE and IgG production. The specific aims of the proposed research are:

1. Determination of the effect of anti-IgE therapy on FcεRI expression and basophil responses. We will first confirm that anti-IgE therapy causes a reduction in the FcεRI level on basophils and then analyze whether this occurs at a transcriptional level. We will confirm that the therapy causes a reduction in basophil response to cross-linkage of FcεRI and then determine whether it also affects basophil response induced by non-IgE stimuli. The effect of the therapy on the FcεRI level on skin mast cells will also be investigated.
2. Determination of the effect of anti-IgE therapy on FcεRII expression and antigen presentation. We will determine whether the therapy results in a down-regulation of FcεRII/CD23 on B cells. Because of the demonstrated function of FcεRII/CD23 in antigen presentation, we will determine the antigen presentation to T cells by B cells from anti-IgE-treated and control subjects.
3. Determination of the effect of anti-IgE therapy on antibody production. We will determine whether anti-IgE therapy results in a suppression of IgE production, in addition to sequestration of IgE. Whether IgE-anti-IgE complexes directly suppress IgE production by B cells in vitro will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Mild or moderate persistent asthma
* Allergic rhinitis
* Atopic dermatitis

Exclusion Criteria:

* Other lung diseases
* Blood clotting disorder
* Pregnant or lactating women

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2004-02; Primary Completion 2012-10-17 (Actual); Study Completion 2012-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fu-Tong Liu, M.D., Ph.D., Principal Investigator — University of California, Davis
Locations (1):
- UC Davis Department of Dermatology, Sacramento, California, United States

REFERENCES:
- See also: University of California-Davis Department of Dermatology Clinical Research — http://www.ucdmc.ucdavis.edu/dermatology/research/clinical

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Omalizumab | Placebo
Started | 3 | 3
First Intervention | 3 | 3
Second Intervention | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omalizumab | Placebo | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 5
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: FcεRI (High Affinity Receptor) Levels at 3 Months
Description: Skin biopsies were collected from patients after 0 (pre), 3 (pos1) and 6 (pos2) months of omalizumab (P11, P36, P42) or placebo (P7 and P38) treatment. The skin was fixed and the paraffin-embedded sections were stained for high affinity receptors. The average numbers of positively stained cells in each field were counted under a microscope at 400X magnification.
Time Frame: 3 months
Population: Skin biopsy was not collected from one of the subjects randomized to placebo.
Measure: Mean (Full Range); unit: Positive cells per field
Groups:
- Omalizumab: The subjects will be randomized to a treatment group and a placebo group. Prior to Omalizumab administration, all subjects will undergo screening studies, including spirometry, blood test and skin test. Blood test includes comprehensive metabolic panel, CBC, and total and free IgE levels. Skin test will be done with a panel of 7 common allergens.
- Placebo: The subjects will be randomized to a treatment group and a placebo group. Prior to placebo administration, all subjects will undergo screening studies, including spirometry, blood test and skin test. Blood test includes comprehensive metabolic panel, CBC, and total and free IgE levels. Skin test will be done with a panel of 7 common allergens.
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 3 | 2
Positive cells per field | 20.5 [3 to 38] | 13.66 [8 to 28]

2. Primary Outcome: FcεRI (High Affinity Receptor) Levels at 6 Months
Description: as for outcome 1
Time Frame: 6 months
Measure: Mean (Full Range); unit: Positive cells per field
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 3 | 2
Positive cells per field | 17 [5 to 38] | 22.5 [15 to 30]

3. Secondary Outcome: Total Sera IgE Levels at 6 Months
Description: Total sera IgE levels are increased upon anti-IgE treatment. Sera from each patient were collected every month after omalizumab (P11, P36 and P42) or placebo (P7, P37 and P38) treatment. The sera IgE levels were measured by ELISA using polyclonal goat anti-human IgE as the capture antibody and HRP-goat anti-human IgE as the detection antibody.
Time Frame: 6 months
Measure: Mean (Full Range); unit: U/ml
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 3 | 3
U/ml | 300 [0 to 600] | 883.33 [300 to 1200]

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Omalizumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3

LIMITATIONS AND CAVEATS:
There are no limitations and caveats.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No